CLINICAL TRIAL: NCT05060718
Title: HONEST-PREPS: Hospital Network Study - Preparation for a Randomized Evaluation of Anti-Pneumonia Strategies
Brief Title: HOspital NEtwork STudy - Preparation for a Randomized Evaluation of Anti-Pneumonia Strategies
Acronym: HONEST-PREPS
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Collaborators: Universiteit Antwerpen (Other); University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, MJM Bonten, Professor of molecular epidemiology of infectious diseases, head of department of medical microbiology, UMC Utrecht
Other Study IDs: HONEST-PREPS
Record Dates: First submitted 2021-07-20; First posted 2021-09-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2022-12

CONDITIONS: Hospital-acquired Pneumonia; Ventilator Associated Pneumonia
MeSH Terms: conditions — Healthcare-Associated Pneumonia; Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hospital Acquired and Ventilator Associated Pneumonia (HAP/VAP) pose a significant burden to patients admitted to the Intensive Care Unit (ICU). Reported incidence ranges from 10-16% in all ICU patients (including HAP and VAP) and around 20-30% in ventilated patients (VAP). Patients with HAP/VAP have a high mortality rate. The estimated attributable mortality of VAP is 6-13%.

Randomized Controlled Trials (RCTs) are the gold standard for evaluating medical interventions, but are difficult to perform in this population. Several preventive and therapeutic treatment options are being developed that will require evaluation in phase-III trials. These trials are challenging due to the relatively low incidence of the outcome (e.g. HAP/VAP) or of the domain under study (e.g. specific antibiotic resistant infections) and the requirement of informed consent in critically ill patients. There is a need for a well-organized and well-trained international RCT network that enables efficient execution of a series of RCTs in this population.

The aim of the current study is to set up an infrastructure to prospectively enroll patients at risk of HAP/VAP in ICUs in several European countries. Site personnel will be trained to obtain a GCP (Good Clinical Practice) certification (if not already done), to timely identify and enroll patients at risk of HAP/VAP, to timely identify occurrence of HAP/VAP, collect informed consent forms, collect source data, enter data into a clinical database, and use a dedicated system to reply to queries. Site sample collection, processing, identifying the causative organism, and antibiotic susceptibility testing will be validated and adapted if required where possible. Where site infrastructure and regulations allow, the possibility of automated data collection of included participants will be explored to ensure sustainability of the future platform. Furthermore, collected data will be used to inform future diagnostic, preventive and therapeutic trials. E.g. they may support assumptions in sample size calculations and expected number of enrolled participants, they may help in prioritizing interventions, or they may be used in simulations of adaptive trials to optimize decision rules.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* At risk of acquiring bacterial HAP or VAP during ICU stay, defined as meeting all of the following criteria:

  * expected or documented hospital length of stay of more than 48 hours
  * admitted to the ICU

Exclusion Criteria:

* Death is deemed to be imminent or inevitable during this hospital admission AND one or more of the patient, substitute decision maker or attending physician are not committed to full active treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to an ICU at risk of bacterial HAP/VAP are eligible to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 2165 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
To determine the quality and efficiency of a research platform for HAP/VAP in ICUs by measuring the timeliness of enrolling eligible patients. | Through study completion, an average of 2 years
  Assess the proportion of screened, eligible patients at risk of developing HAP or VAP by being enrolled within 48 hours of ICU admission.
To determine the quality and efficiency of a research platform for HAP/VAP in ICUs by capturing bacterial HAP/VAP episodes. | Through study completion, an average of 2 years
  Analyse the proportion of enrolled patients who develop HAP/VAP during the initial ICU admission and who are registered in the eCRF (electronic Case Report Form) within 24 hours after onset. Onset is defined as the time of X-ray showing an infiltrate confirming HAP/VAP for patients meeting HAP/VAP FDA criteria.

SECONDARY OUTCOMES:
To determine the incidence of HAP/VAP at the ICU. | From the date of enrolment through to the date of ICU discharge, an average of 11 days
  -Incidence of HAP and VAP per 1,000 patient-days
To determine the implementation of infection prevention and control measures in routine ICU care for prevention of HAP/VAP. | From the date of enrolment through to the date of ICU discharge, an average of 11 days
  -Implementation of ICU-level HAP/VAP infection prevention measures
To determine microbiological etiology of HAP/VAP at the ICU (1). | Between days 7 and 10 after HAP/VAP onset
  -Microbiological cure between 7 and 10 days after HAP/VAP onset (%). (Proportion of patients with positive HAP/VAP diagnosis with the resolution of the symptoms between day 7-10 after the onset)
To determine microbiological etiology of HAP/VAP at the ICU (2). | +/- 48 hours of HAP/VAP onset
  -Distribution of bacterial pathogens (%). (Proportion of identified bacterial pathogens associated with HAP/VAP episode).
To determine microbiological etiology of HAP/VAP at the ICU (3) | +/- 48 hours of HAP/VAP onset
  -Resistance profiles of bacterial pathogens (% resistant) (proportion of resistant bacterial pathogen associated with HAP/VAP episode).
To determine management of HAP/VAP at the ICU (1) | From the date of enrolment through to the date of ICU discharge, on average of 6 days
  -IMV (Invasive Mechanical Ventilation)-free-days up to 28 days after VAP onset (days).
To determine management of HAP/VAP at the ICU (2) | From the date of enrolment through to the date of ICU discharge, on average of 11 days
  -Antibiotic consumption before and after HAP/VAP (type of antibiotic administered per patient).
To determine management of HAP/VAP at the ICU (3). | 90 days after HAP/VAP onset
  -Survival up to 90 days post HAP/VAP onset rate (%) (Proportion of patient's confirmed alive vs. dead in %)
To determine outcome of HAP/VAP at the ICU (1). | From the date of HAP/VAP onset through to the date of ICU discharge, on average of 11 days
  -ICU survival rate (%). (Proportion of patients discharged from ICU alive vs. patients with in-ICU death)
To determine outcome of HAP/VAP at the ICU (2). | From the date of HAP/VAP onset through to the date of hospital discharge, on average of 12 days
  -Hospital survival rate (%). (Proportion of patients discharged from hospital alive vs. patients with in-hospital death)
To determine outcome of HAP/VAP at the ICU (3). | From the date of enrolment through to the date of ICU discharge, on average of 11 days
  -Length of ICU stay before and after HAP/VAP (number of days spent in ICU before and after HAP/VAP onset)
To determine outcome of HAP/VAP at the ICU (4). | From the date of enrolment through to the date of hospital discharge, on average of 12 days
  -Length of hospital stay before and after HAP/VAP (number of days spent in hospital before and after HAP/VAP onset).

CONTACTS AND LOCATIONS:
Overall Officials: Marc Bonten, MD, PhD, Principal Investigator — UMC Utrecht
Locations (16):
- University Trauma Hospital, Tirana, Albania
- Croatia (2):
  - Clinical Hospital Center Rijeka, Rijeka
  - General Hospital Dr Josip Bencevic Slavonski Brod, Slavonski Brod
- Czechia (4):
  - Regional Hospital Kolin, Kolín
  - General University Hospital Prague, Prague
  - University Hospital Kralovske Vinohrady, Prague
  - University Hospital Motol, Prague
- CHU de Limoges, Limoges, France
- Latvia (2):
  - Liepaja Regional Hospital, Liepāja
  - Paul Stradins Clinical University Hospital, Riga
- Romania (2):
  - Central Military Emergency University Hospital "Dr. Carol Davila ", Bucharest
  - Elias University Emergency Hospital, Bucharest
- Serbia (4):
  - Clinical Center of Serbia, Belgrade
  - Clinical Center Kragujevac, Kragujevac
  - Clinical Center of Vojvodina, Novi Sad
  - Institute for Pulmonary Diseases of Vojvodina, Novi Sad

REFERENCES:
- See also: COMBACTE (COMbatting BACterial resistance in Europe) consortium website: HONEST-PREPS is WP2-4 (Work Package) of COMBACTE-NET — https://www.combacte.com/trials/honest-preps/